# Official Protocol Title: Evaluating Local and Regional Immune Responses to Intravesical BCG administration to Patients with Invasive Bladder Cancer

Protocol #: HSC20140002H

Version: 4.0

IRB Approval Date: January, 23. 2017

NCT number: NCT02365207

# **TABLE of Contents**

| STUDY SCHEMA | 3 |
|------------------------------------------------------|----|
| 1.0 OBJECTIVES | 4 |
| 2.0 BACKGROUND | 4 |
| 3.0 DRUG INFORMATION | 5 |
| 4.0 STAGING CRITERIA | 10 |
| 5.0 ELIGIBILITY CRITERIA | 11 |
| 6.0 STUDY PLAN | |
| 7.0 STUDY CALENDAR | 15 |
| 8.0 CRITERIA FOR EVALUATION AND ENDPOINT DEFINITIONS | 15 |
| 9.0 STATISTICAL CONSIDERATIONS | |
| 10.0 REGISTRATION GUIDELINES | |
| 11.0 ETHICAL AND REGULATORY CONSIDERATIONS | 16 |
| 12.0 DATA SAFETY MONITORING | 16 |
| REFERENCES | 20 |

# **Principle Investigator:**

Robert S. Svatek, MD, MSCI Department of Urology
Division of Urologic Oncology
University of Texas Health Science Center San Antonio

Office: 210-567-5676 Fax: 210-567-8095

Email: Svatek@uthscsa.edu

# Co-investigators:

Tyler Curiel, MD **Department of Medicine and Cancer Immunology** University of Texas Health Science Center San Antonio Office: 210 450 5882

Email: curielt@uthscsa.edu

# Study Schema

Patient with known invasive (≥ T1) bladder cancer diagnosed

# Visit 1

Informed Consent;
Research blood/urine
(optional); Symptoms
Questionnaires
(Visit 1 may occur on same
day as BCG week 1)

Neoadjuvant Intravesical BCG (weekly for approximately 3 to 6 weeks);

Symptoms questionnaire weekly; Research urine before and after each BCG instillation

Radical Cystectomy
Research blood, urine, and
tissue, tissue blocks

Post Cystectomy Routine Follow-up (within 90 days postsurgery); Research blood

# 1.0 Objectives

- 1.1 The primary objectives of the study are to determine:
  - a. the ability of intravesical BCG immunotherapy to enhance tumor-specific immunity as measured by autologous T cells proliferation following co-culture with autologous monocyte-derived dendritic cells pulsed with autologous tumor lysate
- 1.2 Secondary objectives of the study are to determine:
  - a. the immune effects of BCG in the tumor microenvironment and tumor-draining lymph nodes
  - b. the extent to which BCG is processed and presented by tumors cells and/or antigenpresenting cells
  - c. the ability of BCG to elicit tumor necrosis/apoptosis in invasive disease
  - d. the pathologic stage of disease following BCG treatment
  - to determine if immune changes elicited by BCG in patients with bladder cancer will
    provide an opportunity for benefit from mTOR inhibition in tumor milieu

# 2.0 Background

# 2.1 Overview

Urothelial carcinoma of the bladder (UCB) accounted for 70,530 new cases of cancer and 14,680 cancer-related deaths in the United States during 2010<sup>1</sup>. Of these new cases, approximately 25% presented as invasive tumors involving the muscular wall of the bladder. Transurethral resection of bladder tumor (TURBT) is an endoscopic procedure that allows for histopathologic assessment and disease staging. TURBT is the primary diagnostic procedure for new and recurrent bladder tumors. TURBT can also be therapeutic for small or non-muscle invasive tumors. However, when muscle-invasive disease is detected, the standard of care involves bladder removal or radical cystectomy (RC) and urinary diversion.

Despite aggressive surgical treatment with bladder removal, up to 50% of patients undergoing RC will experience disease recurrence<sup>2,3</sup>. Chemotherapy given both before and after surgery has been investigated to improve survival for these patients<sup>4-10</sup>. Neoadjuvant chemotherapy renders only a modest improvement in survival- approximately 5-7% absolute benefit in 5-year recurrence free survival<sup>4,11</sup>. Nevertheless neoadjuvant chemotherapy has not been widely adopted due to concerns of toxicity for a modest benefit<sup>11</sup>. In addition, many consider that giving adjuvant chemotherapy for only those patients with high risk pathologic features is a better alternative than treating all patients with neoadjuvant chemotherapy<sup>11</sup>. Current research efforts, therefore, are aimed towards identifying less toxic regimens for use in the neoadjuvant setting. Such effective therapies, especially using those agents with low to moderate toxicity that are easily administered, would be a significant advance in the treatment of invasive bladder cancer. The development of novel, effective therapies, remains an area of unmet need.

# 2.2 <u>Pre-surgical trial</u>

Pre-surgical drug testing is an excellent venue in which paired tumor tissue can be evaluated before and after exposure to a drug to address target specificity, drug delivery, physiologic effects on tumor growth and apoptosis, and correlation of biomarkers with clinical activity<sup>12-15</sup>. Pre-surgical trials have been conducted in radical cystectomy populations were patients were given drugs for 4-7 weeks prior to surgery<sup>12,13</sup>. This approach has been acceptable given the evidence that delaying cystectomy for more than 3 months is not associated with a worse clinical outcome<sup>16-18</sup>. In our protocol, we will seek to characterize the immune effects of intravesical administration in patients undergoing radical cystectomy to help elucidate the anticancer immune mechanisms of BCG in patients with bladder cancer.

#### 2.3 BCG immunotherapy

BCG immunotherapy is the mainstay treatment for high-risk non-muscle invasive bladder cancer. BCG specifically, and Mycobacteria generally, have long been known to be potent immune stimulators but the mechanism of action of BCG in cancer remains incompletely understood. BCG reduces bladder cancer relapse by 50%<sup>19-21</sup> and without it, the risk for cancer relapse is extremely

high (45-80% in non-muscle invasive disease) $^{22-24}$ . In animal models, it has been established that BCG could be effective to treat bladder cancer through immune mechanisms mediating anti-cancer immunity against other cancers, including T cells $^{25}$ , NK cells $^{26}$  and IFN- $\gamma^{27}$ . Nevertheless, many mechanistic details are lacking, notably to what extent BCG generates BCG-specific and tumor-specific immunity and whether BCG affects tumor tolerance. Recently, it was demonstrated that BCG efficacy is mediated, at least in part, through stimulation and recruitment of T cells into peritumoral draining lymph nodes $^{28}$ . This finding has important implications for the utilization of BCG as discussed below.

Currently BCG is principally used to manage non-muscle invasive bladder cancer and has not been employed to treat muscle-invasive disease, since muscle-invasive disease requires bladder removal. However, to date, BCG is the most immunostimulant utilized in bladder cancer there is increasing evidence that BCG could improve tumor-specific immunity<sup>28,29</sup>. If BCG can improve tumor-specific immunity, then it could be used as an adjuvant therapy in the management of bladder cancers of all stages, including muscle-invasive disease. For example, BCG given to patients with muscle-invasive disease prior to cystectomy could improve tumor-specific immunity and enable patients to improve tumor clearance in cases of nodal or distant metastasis. By increasing tumor-specific immunity and memory T cell responses, BCG could also enable sustained long-term protection from recurrent disease.

# 2.4 Rapamycin and immune modulation.

mTOR is a protein kinase that regulates cell growth, proliferation, and other key elements of cell survival. Rapamycin (sirolimus) has long been used in combination with immunosuppressive agents to prevent organ allograft rejection. However, there is no published human study of normal subjects that shows that rapamycin alone is immune suppressive<sup>30</sup>. In fact, recent publications specifically looking at rapamycin immune effects demonstrate that rapamycin boosts immunity to infections<sup>31-33</sup>, accelerates memory CD8<sup>+</sup> T cell differentiation<sup>33</sup>, and improves antigen-specific immunity<sup>33</sup>. Further, rapamycin fed to mice prolongs lifespan<sup>34</sup>, which is inconsistent with significant immunosuppression. Finally, immune modulating properties of mTOR inhibition include effects on T cells, interferon (IFN)-γ and other immune mediators critical to anti-cancer immune defenses<sup>33,35-38</sup>. In preclinical studies, we found rapamycin to improve immune responses and improve the activity of BCG. In secondary objectives, we aim to clarify the effect of BCG in the tumor milieu to determine mTOR inhibition could be beneficial. Specifically, we aim to measure the quantity of regulatory immune activity including PD-1 expression and Treg cells which could negatively influence BCG's activity. If these populations are elevated, mTOR inhibition may be beneficial, as we have observed rapamycin to decrease PD-1 T cells.

#### 3.0 Drug Information (TICE® BCG)

- 3.1 Description: TICE® BCG for intravesical use, is an attenuated, live culture preparation of the Bacillus of Calmette and Guerin (BCG) strain of Mycobacterium bovis. The TICE® strain was developed at the University of Illinois from a strain originated at the Pasteur Institute. The medium in which the BCG organism is grown for preparation of the freeze-dried cake is composed of the following ingredients: glycearin, asparagine, citric acid, potassium phosphate, magnesium sulfate, and iron ammonium citrate. The final preparation prior to freeze drying also contains lactose. The freeze-dried BCG preparation is delivered in glass vials, each containing 1 to 8 x 108 colony forming units (CFU) of TICE® BCG which is equivalent to approximately 50 mg wet weight. Determination of in-vitro potency is achieved through colony counts derived from a serial dilution assay. A single dose consists of 1 reconstituted vial (see DOSAGE AND ADMINISTRATION). For intravesical use the entire vial is reconstituted with sterile saline. TICE® BCG is viable upon reconstitution. No preservatives have been added.
- 3.2 <u>Mechanism of Action:</u> TICE® BCG induces a granulomatous reaction at the local site of administration. Intravesical TICE® BCG has been used as a therapy for, and prophylaxis against, recurrent tumors in patients with carcinoma *in situ* (CIS) of the urinary bladder, and to prevent recurrence of Stage TaT1 papillary tumors of the bladder at high risk of recurrence. The precise mechanism of action is unknown but is thought to be related to immune stimulation and subsequent immune-mediated cytotoxicity.
- 3.3 <u>Toxicology</u>: Symptoms of bladder irritability, related to the inflammatory response induced, are reported in approximately 60% of patients receiving TICE® BCG. The symptoms typically begin 4–6 hours after instillation and last 24–72 hours. The irritative side effects are usually seen following the third instillation, and tend to increase in severity after each administration.

<u>Clinical Studies</u>: To evaluate the efficacy of intravesical administration of TICE® BCG in the treatment of carcinoma in situ, patients were identified who had been treated with TICE® BCG under six different Investigational New Drug (IND) applications in which the most important shared aspect was the use of an induction plus maintenance schedule. Patients received TICE® BCG (50 mg; 1 to 8 x 10<sup>8</sup> CFU) intravesically, once weekly for at least 6 weeks and once monthly thereafter for up to 12 months. A longer maintenance was given in some cases. The study population consisted of 153 patients, 132 males, 19 females, and 2 unidentified as to gender. Thirty patients lacking baseline documentation of CIS and four patients lost to follow-up were not evaluable for treatment response. Therefore, 119 patients were available for efficacy evaluation. The mean age was 69 years (range: 38–97 years). There were two categories of clinical response: (1) Complete Histological Response (CR), defined as complete resolution of carcinoma in situ documented by cystoscopy and cytology, with or without biopsy; and (2) Complete Clinical Response Without Cytology (CRNC), defined as an apparent complete disappearance of tumor upon cystoscopy. The results of a 1987 analysis of the evaluable patients are shown in Table I.

| TABLE I: THE RE | SPONSE OF I | PATIENTS WITH | I CIS BLADDE | R CANCER IN | I SIX IND STUDIES |
|---|---|---|---|---|---|
| | Entered | Evaluable | CR | CRNC | Overall Response |
| No. (%)Of Patients | 153 | 119 (78%) | 54 (46%) | 36 (30%) | 90 (76%) |
| A 1989 update of thes | se data is pres | ented in Table I | . The median o | duration of follo | w-up was 47 months. |

#### TABLE II: FOLLOW-UP RESPONSE OF PATIENTS WITH CIS BLADDER CANCER IN SIX IND STUDIES

| | 1989 Status | of 90 Responders | (CR or CRNC) | |
|------------------|-------------|------------------|---------------|---------|
| | 1987/CR | 1987/CRNC | 1987 Response | |
| Response | n = 54 | n = 36 | n = 90 | Percent |
| CR | 30 | 15 | 45 | 50 |
| CRNC | 0 | 0 | 0 | 0 |
| Unrelated Deaths | 6 | 6 | 12 | 13 |
| Failure | 18 | 15 | 33 | 37 |

There was no significant difference in response rates between patients with or without prior intravesical chemotherapy. The median duration of response, calculated from the Kaplan-Meier curve as median time to recurrence, is estimated at 4 years or greater. The incidence of cystectomy for 90 patients who achieved a complete response (CR or CRNC) was 11%. The median time to cystectomy in patients who achieved a complete response (CR or CRNC) exceeded 74 months. The efficacy of intravesical TICE® BCG in preventing the recurrence of a TaT1 bladder cancer after complete transurethral resection of all papillary tumors was evaluated in two openlabel randomized phase III clinical trials. Initial diagnosis of patients included in the studies was determined by cystoscopic biopsies. One was conducted by the Southwestern Oncology Group (SWOG) in patients at high risk of recurrence<sup>39</sup>. High risk was defined as two occurrences of tumor within 56 weeks, any stage T1 tumor, or three or more tumors presenting simultaneously. The second study was conducted at the Nijmegen University Hospital; Nijmegen, The Netherlands. In this study patients were not selected for high risk of recurrence. In both studies treatment was initiated between 1 and 2 weeks after TUR. In the SWOG trial (study 8795) patients were randomized to TICE® BCG or mitomycin C (MMC)<sup>39</sup>. Both drugs were given intravesically weekly for 6 weeks, at 8 and 12 weeks, and then monthly for a total treatment duration of 1 year. Cystoscopy and urinary cytology were performed every 3 months for 2 years. Patients with progressive disease or residual or recurrent disease at or after the 6 month follow-up were removed from the study and were classified as treatment failures.

A total of 469 patients was entered into the study: 237 to the TICE® BCG arm and 232 to the MMC arm. Twenty-two patients were subsequently found to be ineligible, and 66 patients had concurrent CIS, and were analyzed separately. Four patients were lost to follow-up, leaving 191 evaluable patients in the TICE® BCG arm and 186 in the MMC arm. Of the patients, 84% were male and 16% were female. The average age of these patients was 65 years old. The Kaplan-Meier estimates of 2 year disease-free survival are shown in Table III. The difference in disease-free survival time between the two groups was statistically significant by the log rank test (p=0.03). The 95% confidence interval of the difference in 2 year disease-free survival was  $12\% \pm 10\%$ . No statistically significant differences between the groups were noted in time to tumor progression, tumor invasion, or overall survival.

| TABLE III: RESULTS O | F SWOG STUDY 8795 | |
|---|---|---|
| | TICE® BCG Arm | MMC Arm |
| | N = 191 | N = 186 |
| Estimated Disease-Free Survival at 2 years 95% Confidence Interval (CI) | 57%<br>(50%, 65%) | 45%<br>(38%, 53%) |

In the Nijmegen study, the efficacy of three treatments was compared: TICE substrain BCG, Rijksinstituut voor Volksgezondheid en Milieuhygiene substrain BCG (BCG-RIVM), and MMC. TICE® BCG and BCG-RIVM were given intravesically weekly for 6 weeks. In contrast to the SWOG study, maintenance BCG was not given. Mitomycin C was given intravesically weekly for 4 weeks and then monthly for a total duration of treatment of 6 months. Cystoscopy and urinary cytology were performed every 3 months until recurrence. A total of 469 patients was enrolled and randomized. Thirty-two patients were not evaluable, 17 were ineligible, 15 were withdrawn before treatment, and 50 had concurrent CIS and were analyzed separately, leaving 387 evaluable patients: 117 in the TICE® BCG arm, 134 in the BCG-RIVM arm, and 136 in the MMC arm. Twenty-eight patients (24%) in the TICE® BCG arm, 32 patients (24%) in the BCG-RIVM arm and 24 patients (18%) in the MMC arm had TaG1 tumors. The median duration of follow-up was 22 months (range 3–54 months). The Kaplan-Meier estimates of 2 year disease-free survival are shown in Table IV. The differences in disease-free survival among the three arms were not statistically significant by the log-rank test (p=0.08).

| TABLE IV: RESULTS OF NIJMEGEN STUDY | | | |
|---|---|---|---|
| | TICE® BCG Arm | BCG-RIVM Arm | MMC Arm |
| | N = 117 | N = 134 | N = 136 |
| Estimated Disease-Free Survival at 2 years<br>95% Confidence Interval (CI) | 53%<br>(44%, 64%) | 62%<br>(53%, 72%) | 64%<br>(55%, 74%) |

In both the SWOG 8795 study and the Nijmegen study, acute toxicity was more common, and usually more severe, with TICE® BCG than with MMC (see ADVERSE REACTIONS).

- Warnings: BCG LIVE (TICE® BCG) is not a vaccine for the prevention of cancer. BCG Vaccine, U.S.P., not BCG LIVE (TICE® BCG), should be used for the prevention of tuberculosis. For vaccination use, refer to BCG Vaccine, U.S.P. prescribing information. TICE® BCG is an infectious agent. Physicians using this product should be familiar with the literature on the prevention and treatment of BCG-related complications, and should be prepared in such emergencies to contact an infectious disease specialist with experience in treating the infectious complications of intravesical BCG. The treatment of the infectious complications of BCG requires long-term, multiple-drug antibiotic therapy. Special culture media are required for mycobacteria, and physicians administering intravesical BCG or those caring for these patients should have these media readily available.
- 3.5.1 Instillation of TICE® BCG with an actively bleeding mucosa may promote systemic BCG infection. Treatment should be postponed for at least one week following transurethral resection, biopsy, traumatic catheterization, or gross hematuria.
- 3.5.2 Deaths have been reported as a result of systemic BCG infection and sepsis.2,3 Patients should be monitored for the presence of symptoms and signs of toxicity after each intravesical treatment. Febrile episodes with flu-like symptoms lasting more than 72 hours, fever ≥103°F, systemic manifestations increasing in intensity with repeated instillations, or persistent abnormalities of liver function tests suggest systemic BCG infection and may require antituberculous therapy. Local symptoms (prostatitis, epididymitis, orchitis) lasting more than 2–3 days may also suggest active infection.
- 3.5.3 The use of TICE® BCG may cause tuberculin sensitivity. Since this is a valuable aid in the diagnosis of tuberculosis, it is advisable to determine the tuberculin reactivity by PPD skin testing before treatment.
- 3.5.4 Intravesical instillations of BCG should be postponed during treatment with antibiotics, since antimicrobial therapy may interfere with the effectiveness of TICE® BCG (see PRECAUTIONS). TICE® BCG should not be used in individuals with concurrent infections. Small bladder capacity has been associated with increased risk of severe local reactions and should be considered in deciding to use TICE® BCG therapy.
- **3.6** Management of Serious BCG Complications: Acute, localized irritative toxicities of TICE® BCG may be accompanied by systemic manifestations, consistent with a "flu-like" syndrome. Systemic adverse

effects of 1–2 days' duration such as malaise, fever, and chills often reflect hypersensitivity reactions. However, symptoms such as fever of ≥38.5°C (101.3°F), or acute localized inflammation such as epididymitis, prostatitis, or orchitis persisting longer than 2–3 days suggest active infection, and evaluation for serious infectious complication should be considered.

3.6.1 In patients who develop persistent fever or experience an acute febrile illness consistent with BCG infection, two or more anti-mycobacterial agents should be administered while diagnostic evaluation, including cultures, is conducted and BCG treatment should be discontinued. Negative cultures do not necessarily rule out infection. Physicians using this product should be familiar with the literature on prevention, diagnosis, and treatment of BCG-related complications and, when appropriate, should consult an infectious disease specialist or other physician with experience in the diagnosis and treatment of mycobacterial infections. TICE® BCG is sensitive to the most commonly used antituberculous agents (isoniazid, rifampin and ethambutol). TICE® BCG is not sensitive to pyrazinamide.

#### 3.7 PRECAUTIONS:

- 3.7.1 TICE® BCG contains live mycobacteria and should be prepared and handled using aseptic technique (see **Preparation of Agent** subsection of DOSAGE AND ADMINISTRATION). BCG infections have been reported in health care workers preparing BCG for administration. Needle stick injuries should be avoided during the handling and mixing of TICE® BCG. Nosocomial infections have been reported in patients receiving parenteral drugs which were prepared in areas in which BCG was prepared.4
- 3.7.2 BCG is capable of dissemination when administered by intravesical route and serious reactions, including fatal infections, have been reported in patients receiving intravesical BCG.3 Care should be taken not to traumatize the urinary tract or to introduce contaminants into the urinary system. Seven to 14 days should elapse before TICE® BCG is administered following TUR, biopsy, or traumatic catheterization.
- 3.7.3 TICE® BCG should be administered with caution to persons in groups at high risk for HIV infection

#### 3.8 Drug Interactions

- 3.8.1 Drug combinations containing immunosuppressants and/or bone marrow depressants and/or radiation interfere with the development of the immune response and should not be used in combination with TICE® BCG. Antimicrobial therapy for other infections may interfere with the effectiveness of TICE® BCG. There are no data to suggest that the acute, local urinary tract toxicity common with BCG is due to mycobacterial infection and antituberculosis drugs (e.g., isoniazid) should not be used to prevent or treat the local, irritative toxicities of TICE® BCG.
- 3.8.2 <u>Carcinogenesis, Mutagenesis, Impairment of Fertility:</u> TICE® BCG has not been evaluated for its carcinogenic, mutagenic potentials or impairment of fertility.

# 3.9 Pregnancy

- 3.9.1 Teratogenic Effects Pregnancy Category C: Animal reproduction studies have not been conducted with TICE® BCG. It is also not known whether TICE® BCG can cause fetal harm when administered to a pregnant woman or can affect reproductive capacity. TICE® BCG should not be given to a pregnant woman except when clearly needed. Women should be advised not to become pregnant while on therapy.
- 3.10 <u>Nursing Mothers:</u>It is not known whether TICE® BCG is excreted in human milk. Because many drugs are excreted in human milk and because of the potential for serious adverse reactions from TICE® BCG in nursing infants, it is advisable to discontinue nursing or to discontinue the drug, taking into account the importance of the drug to the mother.
- 3.11 <u>Pediatric Use:</u> Safety and effectiveness of TICE® BCG for the treatment of superficial bladder cancer in pediatric patients have not been established.
- 3.12 Geriatric Use: Of the total number of subjects in clinical studies of TICE® BCG, the average age was 66 years old. No overall difference in safety or effectiveness was observed between older and younger subjects. Other reported clinical experience has not identified differences in response between elderly and younger patients, but greater sensitivity of some older individuals to BCG cannot be ruled out.

# 3.13 ADVERSE REACTIONS

Symptoms of bladder irritability, related to the inflammatory response induced, are reported in approximately 60% of patients receiving TICE® BCG. The symptoms typically begin 4–6 hours after instillation and last 24–72 hours. The irritative side effects are usually seen following the third instillation, and tend to increase in severity after each administration.

The irritative bladder adverse effects can usually be managed symptomatically with products such as

pyridium, propantheline bromide, oxybutynin chloride and acetaminophen. The mechanism of action of the irritative side effects has not been firmly established, but is most consistent with an immunological mechanism.3 There is no evidence that dose reduction or antituberculous drug therapy can prevent or lessen the irritative toxicity of TICE® BCG. "Flu-like" symptoms (malaise, fever, and chills) which may accompany the localized, irritative toxicities often reflect hypersensitivity reactions which can be treated symptomatically. Antihistamines have also been used.5 Adverse reactions to TICE® BCG tend to be progressive in frequency and severity with subsequent instillation. Delay or postponement of subsequent treatment may or may not reduce the severity of a reaction during subsequent instillation. Although uncommon, serious infectious complications of intravesical BCG have been reported.2,3,6 The most serious infectious complication of BCG is disseminated sepsis with associated mortality. In addition, M. bovis infections have been reported in lung, liver, bone, bone marrow, kidney, regional lymph nodes, and prostate in patients who have received intravesical BCG. Some male genitourinary tract infections (orchitis/epididymitis) have been resistant to multiple drug antituberculous therapy and required orchiectomy. If a patient develops persistent fever or experiences an acute febrile illness consistent with BCG infection, BCG treatment should be discontinued and the patient immediately evaluated and treated for systemic infection (see WARNINGS). The local and systemic adverse reactions reported in a review of 674 patients with

| TABLE V: SUMMARY OF ADVERSE EFFECTS SEEN IN 674 PATIENTS WITH | |
|------------------------------------------------------------------|---|
| SUPERFICIAL BLADDER CANCER, INCLUDING 153 WITH CARCINOMA IN SITU | J |

| Percent of Patients | | | Percen | Percent of Patients | |
|---|---|---|---|---|---|
| Adverse<br>Event | N | Overall<br>(Grade ≥3) | Adverse<br>Event | N | Overall<br>(Grade ≥3) |
| Dysuria | 401 | 60% (11%) | Arthritis/Myalgia | 18 | 3% (<1%) |
| Urinary Frequency | 272 | 40% (7%) | Headache/Dizziness | 16 | 2% (0) |
| Flu-Like Syndrome | 224 | 33% (9%) | Urinary Incontinence | 16 | 2% (0) |
| Hematuria | 175 | 26% (7%) | Anorexia/Weight Loss | 15 | 2% (<1%) |
| Fever | 134 | 20% (8%) | Urinary Debris | 15 | 2% (<1%) |
| Malaise/Fatigue | 50 | 7% (0) | Allergy | 14 | 2% (<1%) |
| Cystitis | 40 | 6% (2%) | Cardiac (Unclassified) | 13 | 2% (1%) |
| Urgency | 39 | 6% (1%) | Genital Inflammation/ | | |
| Nocturia | 30 | 5% (1%) | Abscess | 12 | 2% (<1%) |
| Cramps/Pain | 27 | 4% (1%) | Respiratory (Unclassified) | 11 | 2% (<1%) |
| Rigors | 22 | 3% (1%) | Urinary Tract Infection | 10 | 2% (1%) |
| Nausea/Vomiting | 20 | 3% (<1%) | Abdominal Pain | 10 | 2% (1%) |

TABLE VI: MOST COMMON ADVERSE REACTIONS IN SWOG STUDY 8795\*
Study Arm

| | TICE® BCG | (N = 222) | MMC (N | I = 220) |
|----------------------|------------|-----------|------------|----------|
| Adverse Event | All Grades | Grade ≥3 | All Grades | Grade ≥3 |
| Dysuria | 115 (52%) | 6 (3%) | 77 (35%) | 5 (2%) |
| Urgency/Frequency | 112 (50%) | 5 (2%) | 63 (29%) | 7 (3%) |
| Hematuria | 85 (38%) | 6 (3%) | 56 (25%) | 5 (2%) |
| Flu-Like Symptoms | 54 (24%) | 1 (<1%) | 29 (13%) | 0 |
| Fever | 37 (17%) | 1 (<1%) | 7 (3%) | 0 |
| Pain (Not Specified) | 37 (17%) | 4 (2%) | 22 (10%) | 1 (<1%) |
| Hemorrhagic Cystitis | 19 (9%) | 3 (1%) | 10 (5%) | 0 |
| Chills | 19 (9%) | 0 | 2 (1%) | 0 |
| Bladder Cramps | 18 (8%) | 0 | 9 (4%) | 0 |
| Nausea | 16 (7%) | 0 | 12 (5%) | 0 |
| Incontinence | 8 (4%) | 0 | 3 (1%) | 0 |
| Myalgia/Arthralgia | 7 (3%) | 0 | 0 | 0 |
| Diaphoresis | 7 (3%) | 0 | 1 (<1%) | 0 |
| Rash | 6 (3%) | 1 (<1%) | 16 (7%) | 2 (1%) |

3.14 **OVERDOSAGE** Overdosage occurs if more than one vial of TICE® BCG is administered per instillation. If overdosage occurs, the patient should be closely monitored for signs of active local or systemic BCG infection. For acute local or systemic reactions suggesting active infection, an infectious disease specialist experienced in BCG complications should be consulted.

#### 3.15 DOSAGE AND ADMINISTRATION

The dose for the intravesical treatment of carcinoma *in situ* and for the prophylaxis of recurrent papillary tumors consists of one vial of TICE® BCG suspended in 50 ml preservative-free saline.

#### 3.16 Preparation of Agent

The preparation of the TICE® BCG suspension should be done using aseptic technique. To avoid cross-contamination, parenteral drugs should not be prepared in areas where BCG has been prepared. A separate area for the preparation of the TICE® BCG suspension is recommended. All equipment, supplies and receptacles in contact with TICE® BCG should be handled and disposed of as biohazardous. The pharmacist or individual responsible for mixing the agent should wear gloves and take precautions to avoid contact of BCG with broken skin. If preparation cannot be performed in a biocontainment hood, then a mask and gown should be worn to avoid inhalation of BCG organisms and inadvertent exposure to broken skin. Option-1 (Using Syringe Method)

Draw 1 ml of sterile, preservative-free saline (0.9% Sodium Chloride Injection U.S.P.) at 4–25°C, into a small syringe (e.g., 3 ml) and add to one vial of TICE® BCG to resuspend. Gently swirl the vial until a homogenous suspension is obtained. Avoid forceful agitation which may cause clumping of the mycobacteria. Dispense the cloudy TICE® BCG suspension into the top end of a catheter-tip syringe which contains 49 ml of saline diluent, bringing the total volume to 50 ml. To mix, gently rotate the syringe. Option-2 (Using Reconstitution Accessories)

Reconstitution Accessories may be provided with each TICE® BCG product order. Please refer to the Instructions For Use provided with the accessories for a full description of the product reconstitution procedures using these accessories.

The reconstituted TICE® BCG should be kept refrigerated (2–8°C), protected from exposure to direct sunlight, and used within 2 hours. Unused solution should be discarded after 2 hours.

**Note:** DO NOT filter the contents of the TICE® BCG vial. Precautions should be taken to avoid exposing the TICE® BCG to direct sunlight. Bacteriostatic solutions must be avoided. In addition, use only sterile preservative-free saline, 0.9% Sodium Chloride Injection U.S.P. as diluent.

#### 3.17 HOW SUPPLIED

TICE® BCG is supplied in a box of one vial of TICE® BCG. Each vial contains 1 to 8 x 108 CFU, which is equivalent to approximately 50 mg (wet weight), as lyophilized (freeze-dried) powder. NDC 0052-0602-02.

# 3.18 STORAGE

The intact vials of TICE® BCG should be stored refrigerated, at 2–8°C (36–46°F).

This agent contains live bacteria and should be protected from **direct** sunlight. The product should not be used after the expiration date printed on the label.

# 4.0 Staging Criteria

# Bladder cancer Primary Tumor (T)

# Clinical Stage

- cT1 Invades subepithelial connective tissue (lamina propria)
- cT2 Muscle-invasive
- cT3 Residual mass on exam under anesthesia following TURBT
- cT4 Clinically fixed disease on exam under anesthesia

# Pathologic Stage

- pT1 Invades subepithelial connective tissue (lamina propria)
- pT2 Muscle-invasive
- pT3 Invades perivesicle fat
- pT4 Invades adjacent organs (prostate, vagina, uterus, bone, etc...)

# Histiologic subtypes

Urothelial cell carcinoma (Transitional cell carcinoma) Squamous cell carcinoma Adenocarcinoma or glandular carcinoma

# Sarcomatoid carcinoma Micropapillary carcinoma

#### Histiologic grade

High-grade Poorly- or un-differentiated

# 5.0 Eligibility Criteria

#### Inclusion Criteria:

- 5.1 Have suspected or known invasive (≥T1) bladder cancer
- 5.2 Not be in an immunosuppressed state (e.g. HIV +, use of chronic steroids (>1 month))
- 5.3 Be able to give informed consent
- 5.4 Be age 18 or older

#### **Exclusion Criteria:**

- 5.1.1 Have non-invasive (<T1) bladder cancer
- 5.1.2 Is in an immunosuppressed state (e.g. HIV +, use of chronic steroids (>1 month))
- 5.1.3 Unable to give informed consent
- 5.1.4 < 18 or older

# 6.0 Study Plan

#### 6.0 Study Design

This is a one-arm, open label, interventional study. For the purposes of enrollment "study procedure" refers to intravesical BCG instillation. See below for a description of study procedure.

# 6.1 Recruitment

Participants will be recruited through the urology outpatient clinics at the Medical Arts and Research Center (MARC). Attending physicians in the Department of Urology, and selected other personnel who also serve as research staff for this study, will identify prospective study participants. To eliminate selection bias, any patient who presents with invasive bladder cancer and meets the inclusion/exclusion criteria will be given an option to participate in the study. The inclusion of participants or refusal to participate by patients eligible for this study will in no way compromise the quality of health care they will receive.

**Study eligibility** will be determined by investigators and study staff with legitimate access to patient PHI due to their clinical role and/or as members of the research team. Patients who meet the eligibility criteria will be approached by one of the investigators or other members of the study staff to determine whether they are willing to participate in the study. Prior to study entry, the study staff will explain to each potential subject the research objectives, risks and benefits of study participation, alternative treatments available, and the subjects' rights and responsibilities. If the patient agrees to participate, informed consent will be obtained. Research blood and urine may be obtained-OPTIONAL (details in 6.2). Baseline symptoms questionnaires will be administered.

Patients will be approached in a private consult room located within the GU clinic at the MARC. Usual privacy policy practices will be followed. The study procedures and objectives will be described to them and they will be given a copy of the consent document. Participants will also be given contact information for someone they can call with any questions that may arise.

#### 6.2 Visit 1

Routine medical history and demographics and physical exam will be performed during the visit (standard care).

# 6.2.1 Research blood and urine collection & handling OPTIONAL

Research blood and urine may be collected after signing informed consent (OPTIONAL). Approximately 50 mL or 3.5 tablespoons of blood will be taken from a peripheral vein or an indwelling catheter if present and functional specifically for research studies. Study staff will then provide a urine specimen cup and self-catch instruction to the participant. The participant will be able to do this in the privacy of the clinic restroom.

If collected, research blood and urine specimens will be transported to our lab in the STRF in approved containers by qualified personnel. Additional blood will be collected as needed for initial eligibility screening. Urine will be processed by centrifugation and the supernatant will be stored separately from the pellet. Both blood and urine samples are de-identified in the lab per HIPAA protocol.

Baseline symptoms questionnaires will also be administered.

#### 6.3 Neoadjuvant Intravesical BCG Instillation

Prior to undergoing routine radical cystectomy (standard care), participant will receive 3 to 6 weeks of neoadjuvant intravestical BCG instillation weekly as part of the research study procedure. The instillation will be scheduled roughly one week apart pending on the clinic's and participant's schedules, and also participant's reaction to the BCG instillation. BCG Week 1 may occur on the same day as Visit 1.

Intravesical BCG will be given as the intervention measure for treatment of bladder cancer. In brief, following sterile preparation, a Foley catheter is introduced into the bladder thru the urethral meatus. The BCG is instilled through gravity drainage and held in the bladder for approximately 2 hours. Instructions are provided to the patient regarding the proper disposal of the BCG. The duration of BCG treatment is allowed to fluctuate between 3-6 weeks for two reasons: (1) This allows for flexibility in scheduling participants for radical cystectomy as the time from enrollment to cystectomy would vary based on surgeon and patient preferences and on operative room availability. In this manner, the surgery date can be established first and then duration of treatment would be based on amount of time available between enrollment and cystectomy date. In our experience, this "time period" is usually 4-6 weeks; (2) The number of BCG treatments needed to elicit expected immune responses is not known. In fact the current paradigm of 6 weekly treatments has little scientific justification but was based on a rather arbitrary dosing schedule; (3) Allowing for multiple durations of therapy, could provide us with the opportunity to explore differences in immune responses across different dosing duration regimens.

# 6.3.1 Research Urine Collection and Handling Pre and Post-BCG Instillation (research only)

We will collect a urine sample pre-BCG treatment. We will also collect urine samples post-BCG instillations, specifically the <u>second void</u>, which typically occur 4-6 hours post Intravesical BCG treatment. Participants will be given the following options for collection of urine sample post intravesical BCG treatments:

- a) Participant may remain in the clinic for urine collection -OR-
- b) Participant may leave the clinic with a urine sample collection cup and biohazard bag. Participant will be given specific instruction to collect second void post intravesical BCG therapy, and return the sample to the clinic.

Study team member will work with participant on how post BCG therapy urine will be collected and returned to the team. Post-BCG urine collection will take place at weekly during the 3-6 weeks of intravesical BCG treatments. Urine will be processed by centrifugation and the supernatant will be stored separately from the pellet.

# 6.3.2 Dose Modification and Toxicity

BCG at a dose of 1 to 8 x 10<sup>8</sup> is given intravesically for 2 hours, irrespective of weight or age. This dose was chosen because previous experience and standard care with BCG.

Adjustments (1/2 strength or ¼ strength) are allowed for participants demonstrating poor toleration of treatment as is done in the course of usual standard care.

\*Note: Due to the nationwide shortage of BCG, the entire vial (1 full dose) may not be used for the treatment. Patients may elect to receive BCG treatments at standard of care physician.

BCG treatment may be held by the treating physician for clinical reasons such as active urinary tract infection or gross bleeding from the bladder as per standard care. Regardless of dose or amount of BCG given, patients will be allowed to continue with study procedures.

# 6.3.3 Monitoring during BCG Instillation

At each visit (including baseline) symptom questionnaires will be administered prior to any procedures. The symptom questionnaires will assess irritative LUTS present. If BCG Grade 3 bladder toxicity occurs it will result in postponing combined therapy by 1 week, provided that the patient's symptoms resolved.

Participant-reported side effect questionnaires will be administered prior to each weekly instillation to ascertain the previous instillation's effects. Patients will be monitored in the clinic during instillation of BCG.

Adverse event (AE) monitoring will be assessed at each clinic visit, during BCG treatments, and on the day of cystectomy. Safety will be assessed by a urologist with training in administration of intravesical BCG.

Dose-Limiting Toxicity (DLT) - Dose-limiting toxicity (DLT) is defined as any grade 3 or 4 systemic toxicities or evidence of grade 4 bladder toxicity using the National Cancer Institute common toxicity criteria.

6.4 Research Blood, urine, & tissue collection (research only) at the time of Radical Cystectomy (standard care)

Research blood and urine will be collected at radical cystectomy.. Approximately 50 mL or 3.5 tablespoons of blood will be taken from a peripheral vein or an indwelling catheter if present and functional specifically for research studies. The handling method can be found in Section 6.2.1. Voided urine or urine from an indwelling catheter will be collected.

At the time of radical cystectomy, a section of tumor tissue, normal adjacent bladder tissue, and adjacent lymphatic tissue will be taken for immune studies. A small section of the tissue from the bladder (approximately 5 mm x 5 mm x 5 mm) will be taken. Most patients with muscle invasive tumors have large tumors so taking a small section does not compromise pathologic assessment of stage. This research tissue would be excess tumor and would not compromise the ability of the pathologist to stage or grade the tumor, and poses no additional meaningful risk to the patient. To ensure this we clarify that the tumor tissue taken for research represents a small (10% of the tumor volume or less) component of the tumor. If sufficient excess tumor is not available for research purposes, then no research bladder tissue would be removed. We have experience with such post-treatment tumor acquisition for research in bladder cancer studies here at UTHSCSA. For benign adjacent bladder mucosa, we will also take a small section (approximately 5 mm x 5 mm x 5 mm) of tissue. Normally for lymph node dissections, we typically remove 20-60 lymph nodes during a cystectomy. We will isolate several (2-8) lymph nodes to be used for research purposes. The lymph node will removed and then surgically split in half. One half will be sent for pathologic processing and the other half will be used for research. In this way, we do not compromise the ability to pathologically examine the lymph nodes.

13

We will also obtain the tissue blocks from cystectomy on all subjects from pathology where surgery was done.

# 6.5 Post-Radical Cystectomy Follow-up Visit (standard care)

As per routine care, participants will return to clinic approximately within 90 days following surgery for a follow-up visit. During this visit, research blood will be collected.

Approximately 50 mL or 3.5 tablespoons of blood will be taken from a peripheral vein or an indwelling catheter if present and functional specifically for research studies. The research blood specimens will be transported to our lab in the STRF in approved containers by qualified personnel. The blood sample will be de-identified in the lab per HIPAA protocol.

7.0 Study Calendar

| Study | Visit | BCG | BCG | BCG | BCG | BCG | BCG | Cystectomy | Post |
|---|---|---|---|---|---|---|---|---|---|
| Component/Procedures | 1 | Week | Week | Week | Week | Week | Week | - Joseph - J | Cystectomy |
| | _ | 1 | 2 | 3 | <b>4</b> a | 5a | 6a | | (~within 90 |
| | | (may | | | | | | | days post |
| | | be | | | | | | | cystectomy) |
| | | same | | | | | | | |
| | | day as | | | | | | | |
| | | Visit | | | | | | | |
| | | 1) | | | | | | | |
| Informed Consent | R | | | | | | | | |
| Medical History, | S | | | | | | | | |
| Demographics, Physical | | | | | | | | | |
| Exam | | | | | | | | | |
| Assessment of AEs | | R | R | R | R | R | R | | |
| Urinary symptoms | R | R | R | R | R | R | R | | |
| questionnaires | | | | | | | | | |
| Blood Collection | R* | | | | | | | R | R |
| Urine Collection | R* | R | R | R | R | R | R | R | |
| (pre and post treatment | | | | | | | | | |
| urine collected on BCG | | | | | | | | | |
| weeks) | | | | | | | | | |
| Tissue collection | | | | | | | | R | |
| Tissue blocks from | | | | | | | | R | |
| cystectomy procedure | | | | | | | | | |

<sup>&</sup>quot;R" indicates performed only for research purposes and "S" indicates performed for standard care practice a- Additional BCG treatments beyond week 3 will be given selectively to participants based on time interval between study enrollment and scheduled cystectomy date

# 8.0 <u>Criteria for Evaluation and Endpoint Definitions</u>

- 8.1 The primary end-point is taken as difference in tumor-specific immune response (comparing before and after treatment with BCG). Tumor-specific immune response will be measured using a standard T cell proliferation assay. T cell response to autologous tumor will be measured using a paired analysis by utilizing PBMCs collected before and after BCG therapy. Autologous monocyte-derived dendritic cells (moDCs) and autologous T cells will be co-cultured following pulsation of moDCs with whole tumor lysates.
- 8.2 Secondary endpoints are exploratory and will not be considered for determining sample size. Secondary endpoints include (1) description of tumor infiltrating lymphocyte populations following BCG (examining 3 weeks of treatment versus 4,5, or 6 weeks as available); (2) determination of the presence/absence of BCG in lymph nodes following treatment; (3) examining extent of necrosis/apoptosis in tumor following BCG treatment; (4) pathologic assessment of tumor stage following BCG treatment; (5) characterization of systemic immune populations before treatment, at time of cystectomy,

# 9.0 <u>Statistical Considerations</u>

# 9.1 Sample Size Determination

This is a one-arm open label study of the tumor-specific immune effect of BCG in participants undergoing radical cystectomy for bladder cancer. The sample size calculation is based on one-sided testing on the proportion of subjects who experience an increase in T cell proliferation (≥100% increase in proliferative index during the proliferation assay) in post treatment assessment compared to pretreatment assessment with power=90% and target alpha=5%. The null proportion responding is taken to be 0.10 and the desired proportion responding is specified as greater than or equal to 0.50. The estimated sample size, under these assumptions, is 10. In order to achieve this number

<sup>\*</sup> Optional blood and urine collection

we would need to consent 25 participants to account for completion rate and assay variability.

Sample size calculations were run using Stata 10.1 (College Station, Texas).

#### Data analysis

Descriptive graphs will be developed to describe immune subpopulations and immunodynamic end points on paired samples on an intraindividual basis. For all other immune analyses, comparisons between groups will be conducted using the nonparametric Wilcoxon rank-sum test and comparison within groups will be conducted using the Wilcoxon signed-rank test. Correlation will be analyzed with the Spearman rank test.

# 10.0 Registration Guidelines

Participants will be registered on to IDEAS.

#### 11.0 Ethical and regulatory

The following must be observed to comply with Food and Drug Administration regulations for the conduct and monitoring of clinical investigations; they also represent sound research practice:

#### Informed Consent

The principles of informed consent are described by Federal Regulatory Guidelines (Federal Register Vol. 46, No. 17, January 27, 1981, part 50) and the Office for Protection from Research Risks Reports: Protection of Human Subjects (Code of Federal Regulations 45 CFR 46). They must be followed to comply with FDA regulations for the conduct and monitoring of clinical investigations.

# Institutional Review

This study must be approved by an appropriate institutional review committee as defined by Federal Regulatory Guidelines (Ref. Federal Register Vol. 46, No. 17, January 27, 1981, part 56) and the Office for Protection from Research Risks Reports: Protection of Human Subjects (Code of Federal Regulations 45 CFR 46).

# 12.0 Data and Safety Monitoring Oversight

A Data and Safety Monitoring Plan (DSMP) is required for all an individual protocols conducted at CTRC. All protocols conducted at CTRC are covered under the auspices of the CTRC Institutional Data Safety Monitoring Plan.

The CTRC Institutional DSMP global policies provide individual trials with:

- institutional policies and procedures for institutional data safety and monitoring,
- an institutional guide to follow,
- monitoring of protocol accrual by the CTRC Protocol Review Committee,
- review of study forms and orders by the Forms Committee,
- tools for monitoring safety events,
- monitoring of UPIRSO's by the Director of Quality Assurance and DSMC,
- determining level of risk (Priority of Audit Level Score PALS),
- oversight by the Data Safety Monitoring Committee (DSMC), and
- verification of protocol adherence via annual audit for all Investigator Initiated Studies by the CTRC Quality Assurance Division.

#### Monitoring Safety:

Due to the low risk associated with participation in this protocol, the Principal Investigator will perform primary assessment of adverse events, adverse event trends and treatment effects on this study. The PI will conduct independent review and report findings yearly to the CTRC Data Safety Monitoring Committee (DSMC) and the UTHSCSA IRB.

Baseline events and adverse events will be captured using the CTRC Master Adverse Events Document for each patient using CTCAE V. (specify version you will use in this protocol) for the grading and attribution of adverse events. Usage of the CTRC Master Adverse Events Document centrally documents:

- · the event and grades the seriousness of it,
- if the event was a change from baseline,
- · determines the relationship between the event and study intervention,
- if the event was part of the normal disease process, and
- what actions were taken as a result of the event.

#### Safety Definitions:

For this study, the following safety definitions will be applicable:

Adverse Event Definition: An adverse event (AE) is defined as any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research For this study, all adverse events will be documented starting with specify here when you want to start collecting adverse event information, generally this would be with the first dose of the study drug and ending 30 days after the last dose of study drug is received.

Serious Adverse Event Definition: is any adverse event that:

- 1. results in death;
- 2. is life-threatening (places the subject at immediate risk of death from the event as it occurred);
- 3. results in inpatient hospitalization or prolongation of existing hospitalization;
- 4. results in a persistent or significant disability/incapacity;
- 5. results in a congenital anomaly/birth defect; or
- 6. based upon appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the other outcomes listed in this definition

Unanticipated Problems Involving Risks to Subjects or Others Definition: Unanticipated problem involving risk to subjects or others includes any incident, experience or outcome that meets all of the following criteria:

- A. unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document; and (b) the characteristics of the subject population being studied (note: the unfounded classification of a serious adverse event as "anticipated" constitutes serious non-compliance);
- B. definitely related or probably related to participation in the research; and
- C. suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized

# Reporting Requirements

For this study, all Master Adverse Events Documents collected on participants for this protocol will be reviewed by the Principal Investigator at each study visit/as they occur to determine if a serious safety problem has emerged that result in a change or early termination of a protocol such as:

- dose modification,
- suspending enrollment due to safety or efficacy, or
- termination of the study due to a significant change in risks or benefits.

The PI will use clinical judgment to make dose reduction and dose delay in BCG as per standard of care. Since these adjustments are very patient-specific, this will be done on a case-by-case basis.

As per the CTRC DSMP, any protocol modifications, problematic safety reports, unanticipated problems, and suspension or early termination of a trial must be reported to all members of the research team Suspension and early termination of a trial must also be reported immediately to the Director of Quality Assurance (DQA) who will promptly notify the sponsor and the UTHSCSA IRB.

The PI will review the Master Adverse Events documents to determine the significance of the reported events and will file the Investigator Initiated Study Quarterly DSMC Report Form on a yearly basis with the CTRC DSMC. The Investigator Initiated Study Quarterly DSMC Report Form includes information on adverse events, current dose levels, number of participants enrolled, significant toxicities per the protocol,

patient status (morbidity and mortality), dose adjustments with observed response, and any interim findings. Any trend consisting of three or more of the same event will be reported to the CTRC DSMP for independent review outside of the quarterly reporting cycle, which begins three months following protocol start up. Conflict of interest is avoided by the independent review of the CTRC DSMC and by ongoing independent review of adverse events trends by the Director of Quality Assurance.

All SAE and UPRISO's will be reported following CTRC and UTHSCSA institutional guidelines.

| | | 0 |
|---|---|---|
| UTHSCSA SAE/UPRISO REPORTING REQUIREMENTS | | |
| Type Event | Report to | Timeframe |
| All AE, SAE and UPIRSO | Regulatory Affairs and DOA | Same as other notification timeframes except for SAE/AE which should be reported on Monday for the prior week of PI being made aware |
| All AE, SAE allu UPIRSU | Regulatory Affairs and DQA | for the prior week of Fr being made aware |
| SAE | Clinical Trial Sponsor | within 24 hours of PI being made aware |
| AE/SAE | UTHSCSA IRB | Annually |
| UPIRSO - all | Clinical Trial Sponsor | within 24 hours of the PI determining a UPIRSO exists |
| UPIRSO - life threatening | UTHSCSA IRB | within 48 hours of the PI determining a UPIRSO exists |
| UPIRSO - non-life threatening | UTHSCSA IRB | within 7 days of the PI determining a UPIRSO exists |

Include the following adverse event reporting requirement tables for NCI Trials supported by Grant or Contract Funding:

TABLE A: Expedited Reporting for Phase I Studies (including hospitalization\* to NCI Investigational Drug Branch (IDB)

| UNEXPECTED EVENT | | EXPECTED EVENT | |
|---|---|---|---|
| GRADES 2 - 3 Attribution of Possible, Probable or Definite | GRADES 4 - 5 Regardless of Attribution | GRADES 1 – 3 | GRADES 4 - 5 Regardless of Attribution |
| Grade 2 - Expedited report within 10 working days | Report by phone to IDB within 24 hrs. Expedited report to follow within 10 working days. | Adverse Event Expedited Reporting NOT required. | Report by phone to IDB within 24 hrs. Expedited report to follow within 10 working days. |
| Grade 3 - Report by phone to IDB within 24 hrs. Expedited report to follow within 10 working days. (Grade 1 - Adverse Event Expedited Reporting NOT required.) | This includes all deaths within 30 days of the last dose of treatment with an investigational agent regardless of attribution. Any late death attributed to the agent (possible, probable, or definite) should be reported | | This includes all deaths within 30 days of the last dose of treatment with an investigational agent regardless of attribution. Any late death attributed to the agent (possible, probable, or definite) should be reported |

<sup>\*</sup> For Hospitalization Only — Any medical event equivalent to CTC Grade 3, 4, 5 which precipitated hospitalization (or prolongation of existing hospitalization) must be reported regardless of requirements for Phase of study, expected or unexpected and attribution.

Expedited reporting may not be appropriate for specific expected adverse events for certain later Phase II and Phase III protocols. In those situations the adverse events that will not have expedited reporting must be specified in the text of the approved protocol. An expected Grade 3 event that is definitely related to the investigational agent is only to be reported if the patient is hospitalized using the generic reporting criteria. For instance, in a trial of an investigational agent where Grade 3 diarrhea requiring hospitalization is expected, only diarrhea requiring ICU care (Grade 4) might be designated for expedited reporting.

Serious adverse events on NCI sponsored trials utilizing a commercially available agent (with no IND's involved) will additionally be reported via the FDA's Medwatch program.

# Assuring Compliance with Protocol and Data Accuracy

As with all studies conducted at CTRC, the PI has ultimate responsibility for ensuring protocol compliance, data accuracy/integrity and responding to recommendations that emanate from monitoring activities. (Please write in here any specific monitoring functions such as source verification etc that are either conducted by the sponsor's monitor or newly implemented CTRC monitoring plan –for example, source verification of data will be performed routinely at each visit/as they occur). Protocol compliance, data accuracy and reporting of events is further ensured by an annual audit conducted by the Data Safety Officer, whose audit report is shared with the PI, the research team, and will be reviewed by the CTRC DSMC.

| DSMB #2 (for Solid Tumors) |
|----------------------------|
| Kevin Kelly, MD |
| Ting Lu, MD |
| Wendy Crabbe, PA, MSN, RN |
| Melissa Nashawati, MPA |
| Yuanyuan Liang, PhD |

#### **REFERENCES**

- 1. JEMAL A, SIEGEL R, XU J, WARD E. CANCER STATISTICS, 2010. CA CANCER J CLIN. SEP-OCT 2010;60(5):277-300.
- 2. SONPAVDE G, KHAN MM, SVATEK RS, ET AL. PROGNOSTIC RISK STRATIFICATION OF PATHOLOGICAL STAGE T2N0 BLADDER CANCER AFTER RADICAL CYSTECTOMY. *BJU INT*. SEP 2011;108(5):687-692.
- 3. SVATEK RS, SHARIAT SF, NOVARA G, ET AL. DISCREPANCY BETWEEN CLINICAL AND PATHOLOGICAL STAGE: EXTERNAL VALIDATION OF THE IMPACT ON PROGNOSIS IN AN INTERNATIONAL RADICAL CYSTECTOMY COHORT. *BJU INTERNATIONAL*. MAR 2011;107(6):898-904.
- **4.** GROSSMAN HB, NATALE RB, TANGEN CM, ET AL. NEOADJUVANT CHEMOTHERAPY PLUS CYSTECTOMY COMPARED WITH CYSTECTOMY ALONE FOR LOCALLY ADVANCED BLADDER CANCER. *N ENGL J MED*. AUG 28 2003;349(9):859-866.
- 5. ADJUVANT CHEMOTHERAPY IN INVASIVE BLADDER CANCER: A SYSTEMATIC REVIEW AND META-ANALYSIS OF INDIVIDUAL PATIENT DATA ADVANCED BLADDER CANCER (ABC) META-ANALYSIS COLLABORATION. *EUR UROL.* AUG 2005;48(2):189-199; DISCUSSION 199-201.
- 6. NEOADJUVANT CHEMOTHERAPY IN INVASIVE BLADDER CANCER: UPDATE OF A SYSTEMATIC REVIEW AND META-ANALYSIS OF INDIVIDUAL PATIENT DATA ADVANCED BLADDER CANCER (ABC) META-ANALYSIS COLLABORATION. *EUR UROL.* AUG 2005;48(2):202-205; DISCUSSION 205-206.
- 7. POLLERA CF. [NEOADJUVANT CHEMOTHERAPY: META-ANALYSIS AND INTERPRETATION OF RESULTS IN BLADDER CANCER]. SUPPL TUMORI. JUL-AUG 2004;3(4):S59-61.
- 8. RUGGERI EM. [META-ANALYSIS OF NEOADJUVANT CHEMOTHERAPY IN LOCALLY ADVANCED BLADDER CANCER]. SUPPL TUMORI. JUL-AUG 2004;3(4):S55-56.

- 9. WINQUIST E, KIRCHNER TS, SEGAL R, CHIN J, LUKKA H. NEOADJUVANT CHEMOTHERAPY FOR TRANSITIONAL CELL CARCINOMA OF THE BLADDER: A SYSTEMATIC REVIEW AND META-ANALYSIS. *J UROL.* FEB 2004;171(2 PT 1):561-569.
- **10.** NEOADJUVANT CHEMOTHERAPY IN INVASIVE BLADDER CANCER: A SYSTEMATIC REVIEW AND META-ANALYSIS. *LANCET.* JUN 7 2003;361(9373):1927-1934.
- **11.** BLACK PC, BROWN GA, GROSSMAN HB, DINNEY CP. NEOADJUVANT CHEMOTHERAPY FOR BLADDER CANCER. *WORLD J UROL*. NOV 2006;24(5):531-542.
- 12. CARTHON BC, WOLCHOK JD, YUAN J, ET AL. PREOPERATIVE CTLA-4 BLOCKADE: TOLERABILITY AND IMMUNE MONITORING IN THE SETTING OF A PRESURGICAL CLINICAL TRIAL. *CLIN CANCER RES.* MAY 15 2010;16(10):2861-2871.
- 13. PRUTHI RS, NIELSEN M, HEATHCOTE S, ET AL. A PHASE II TRIAL OF NEOADJUVANT ERLOTINIB IN PATIENTS WITH MUSCLE-INVASIVE BLADDER CANCER UNDERGOING RADICAL CYSTECTOMY: CLINICAL AND PATHOLOGICAL RESULTS. *BJU INT.* AUG 2010;106(3):349-354.
- 14. CHI KN, EISENHAUER E, FAZLI L, ET AL. A PHASE I PHARMACOKINETIC AND PHARMACODYNAMIC STUDY OF OGX-011, A 2'-METHOXYETHYL ANTISENSE OLIGONUCLEOTIDE TO CLUSTERIN, IN PATIENTS WITH LOCALIZED PROSTATE CANCER. *J NATL CANCER INST.* SEP 7 2005;97(17):1287-1296.
- **15.** ARMSTRONG AJ, NETTO GJ, RUDEK MA, ET AL. A PHARMACODYNAMIC STUDY OF RAPAMYCIN IN MEN WITH INTERMEDIATE- TO HIGH-RISK LOCALIZED PROSTATE CANCER. *CLIN CANCER RES.* JUN 1 2010;16(11):3057-3066.
- **16.** AYRES BE, GILLATT D, MCPHAIL S, ET AL. A DELAY IN RADICAL CYSTECTOMY OF >3 MONTHS IS NOT ASSOCIATED WITH A WORSE CLINICAL OUTCOME. *BJU INT.* SEP 2008;102(8):1045.
- 17. FRADET V, KONETY BR. A DELAY IN RADICAL CYSTECTOMY OF >3 MONTHS IS NOT ASSOCIATED WITH A WORSE CLINICAL OUTCOME. *BJU INT.* JAN 2008;101(2):257-258; AUTHOR REPLY 258-259.

- 18. NIELSEN ME, PALAPATTU GS, KARAKIEWICZ PI, ET AL. A DELAY IN RADICAL CYSTECTOMY OF >3 MONTHS IS NOT ASSOCIATED WITH A WORSE CLINICAL OUTCOME. *BJU INT.* NOV 2007;100(5):1015-1020.
- 19. SYLVESTER RJ, VAN DER MA, LAMM DL. INTRAVESICAL BACILLUS CALMETTE-GUERIN REDUCES THE RISK OF PROGRESSION IN PATIENTS WITH SUPERFICIAL BLADDER CANCER: A META-ANALYSIS OF THE PUBLISHED RESULTS OF RANDOMIZED CLINICAL TRIALS. *J UROL.* NOV 2002;168(5):1964-1970.
- 20. SYLVESTER RJ, VAN DER MEIJDEN AP, WITJES JA, KURTH K. BACILLUS CALMETTE-GUERIN VERSUS CHEMOTHERAPY FOR THE INTRAVESICAL TREATMENT OF PATIENTS WITH CARCINOMA IN SITU OF THE BLADDER: A META-ANALYSIS OF THE PUBLISHED RESULTS OF RANDOMIZED CLINICAL TRIALS. J UROL. JUL 2005;174(1):86-91; DISCUSSION 91-82.
- 21. LAMM DL, BLUMENSTEIN BA, CRISSMAN JD, ET AL. MAINTENANCE BACILLUS CALMETTE-GUERIN IMMUNOTHERAPY FOR RECURRENT TA, T1 AND CARCINOMA IN SITU TRANSITIONAL CELL CARCINOMA OF THE BLADDER: A RANDOMIZED SOUTHWEST ONCOLOGY GROUP STUDY. *J UROL*. APR 2000;163(4):1124-1129.
- 22. KREGE S, GIANI G, MEYER R, OTTO T, RUBBEN H. A RANDOMIZED MULTICENTER TRIAL OF ADJUVANT THERAPY IN SUPERFICIAL BLADDER CANCER: TRANSURETHRAL RESECTION ONLY VERSUS TRANSURETHRAL RESECTION PLUS MITOMYCIN C VERSUS TRANSURETHRAL RESECTION PLUS BACILLUS CALMETTE-GUERIN. PARTICIPATING CLINICS. *J UROL.* SEP 1996;156(3):962-966.
- 23. HENEY NM. NATURAL HISTORY OF SUPERFICIAL BLADDER CANCER. PROGNOSTIC FEATURES AND LONG-TERM DISEASE COURSE. *THE UROLOGIC CLINICS OF NORTH AMERICA*. AUG 1992;19(3):429-433.
- **24.** HENEY NM, AHMED S, FLANAGAN MJ, ET AL. SUPERFICIAL BLADDER CANCER: PROGRESSION AND RECURRENCE. *J UROL.* DEC 1983;130(6):1083-1086.
- **25.** BROGHAMMER EL, RATLIFF TL. IMMUNOTHERAPY OF UROLOGIC TUMORS: PRINCIPLES AND PROGRESS. *UROL ONCOL.* MAR-APR 2002;7(2):45-56.
- **26.** BRANDAU S, RIEMENSBERGER J, JACOBSEN M, ET AL. NK CELLS ARE ESSENTIAL FOR EFFECTIVE BCG IMMUNOTHERAPY. *INT J CANCER*. JUN 1 2001;92(5):697-702.

- 27. RIEMENSBERGER J, BOHLE A, BRANDAU S. IFN-GAMMA AND IL-12 BUT NOT IL-10 ARE REQUIRED FOR LOCAL TUMOUR SURVEILLANCE IN A SYNGENEIC MODEL OF ORTHOTOPIC BLADDER CANCER. *CLIN EXP IMMUNOL.* JAN 2002;127(1):20-26.
- 28. BIOT C, RENTSCH CA, GSPONER JR, ET AL. PREEXISTING BCG-SPECIFIC T CELLS IMPROVE INTRAVESICAL IMMUNOTHERAPY FOR BLADDER CANCER. SCI TRANSL MED. JUN 6 2012;4(137):137RA172.
- 29. BREBAN R, BISIAUX A, BIOT C, RENTSCH C, BOUSSO P, ALBERT ML. MATHEMATICAL MODEL OF TUMOR IMMUNOTHERAPY FOR BLADDER CARCINOMA IDENTIFIES THE LIMITATIONS OF THE INNATE IMMUNE RESPONSE. ONCOIMMUNOLOGY. JAN 1 2012;1(1):9-17.
- **30.** FERRER IR, WAGENER ME, ROBERTSON JM, ET AL. CUTTING EDGE: RAPAMYCIN AUGMENTS PATHOGEN-SPECIFIC BUT NOT GRAFT-REACTIVE CD8+ T CELL RESPONSES. *J IMMUNOL.* AUG 15 2010;185(4):2004-2008.
- 31. JAGANNATH C, LINDSEY DR, DHANDAYUTHAPANI S, XU Y, HUNTER RL, JR., EISSA NT. AUTOPHAGY ENHANCES THE EFFICACY OF BCG VACCINE BY INCREASING PEPTIDE PRESENTATION IN MOUSE DENDRITIC CELLS. *NAT MED.* MAR 2009;15(3):267-276.
- 32. VEZYS V, YATES A, CASEY KA, ET AL. MEMORY CD8 T-CELL COMPARTMENT GROWS IN SIZE WITH IMMUNOLOGICAL EXPERIENCE. NATURE. JAN 8 2009;457(7226):196-199.
- 33. ARAKI K, TURNER AP, SHAFFER VO, ET AL. MTOR REGULATES MEMORY CD8 T-CELL DIFFERENTIATION. *NATURE*. JUL 2 2009;460(7251):108-112.
- **34.** HARRISON DE, STRONG R, SHARP ZD, ET AL. RAPAMYCIN FED LATE IN LIFE EXTENDS LIFESPAN IN GENETICALLY HETEROGENEOUS MICE. *NATURE*. JUL 16 2009;460(7253):392-395.
- **35.** DELGOFFE GM, KOLE TP, ZHENG Y, ET AL. THE MTOR KINASE DIFFERENTIALLY REGULATES EFFECTOR AND REGULATORY T CELL LINEAGE COMMITMENT. *IMMUNITY*. JUN 19 2009;30(6):832-844.
- **36.** HAXHINASTO S, MATHIS D, BENOIST C. THE AKT-MTOR AXIS REGULATES DE NOVO DIFFERENTIATION OF CD4+FOXP3+ CELLS. *J EXP MED.* MAR 17 2008;205(3):565-574.

- **37.** WEICHHART T, SAEMANN MD. THE MULTIPLE FACETS OF MTOR IN IMMUNITY. *TRENDS IMMUNOL.* MAY 2009;30(5):218-226.
- **38.** WEICHHART T, COSTANTINO G, POGLITSCH M, ET AL. THE TSC-MTOR SIGNALING PATHWAY REGULATES THE INNATE INFLAMMATORY RESPONSE. *IMMUNITY*. OCT 17 2008;29(4):565-577.
- 39. LAMM DL, BLUMENSTEIN BA, CRISSMAN JD, ET AL. MAINTENANCE BACILLUS CALMETTE-GUERIN IMMUNOTHERAPY FOR RECURRENT TA, T1 AND CARCINOMA IN SITU TRANSITIONAL CELL CARCINOMA OF THE BLADDER: A RANDOMIZED SOUTHWEST ONCOLOGY GROUP STUDY. *J UROL.* APR 2000;163(4):1124-1129.